CLINICAL TRIAL: NCT05609019
Title: Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Activity of SYHX2005 in Patients With Advanced Solid Tumors
Brief Title: A Study Evaluating SYHX2005 in the Treatment of Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYHX2005-CSP-001
Record Dates: First submitted 2022-10-12; First posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SYHX2005 (Experimental): Stage1 dose-escalation: Patients with advanced solid tumors will receive escalating doses of SYHX2005 as monotherapy.
  Stage2 dose-expansion: Patients with advanced solid tumors will receive SYHX2005 monotherapy at recommended dose (1 or 2 ) in Stage 1 (dose escalation) to evaluate the preliminary antitumor activity of SYHX2005.
  Interventions: Drug: SYHX2005

INTERVENTIONS:
Drug: SYHX2005 — Tablets. Take orally.

SUMMARY:
This is a first-in-human study with the SYHX2005 tablet primarily designed to evaluate the safety and tolerability of SYHX2005 at increasing doses in patients with advanced solid tumors and for whom no standard of care exists. The study will be conducted in two parts: Stage1 dose-escalation and Stage2 dose-expansion. In Stage1, patient enrolment will be proceeded according to a "Accelerated Titration + BOIN" design in order to identify the maximum-tolerated dose (MTD) or recommended dose. In Stage2, preliminary efficacy response will be assessed in patients with advanced solid tumors in use of the recommended dose.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18~70 years old (inclusive).
2. Patients with advanced solid tumors diagnosed histologically or cytologically.
3. Could provide tumor tissue sections or agree to take biopsy for central laboratory biomarker detection.
4. At least one measurable lesion according to RECIST v1.1.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
6. Life expectancy of at least 3 months.
7. Adequate organ function.
8. Males and females with reproductive potential must agree to use medically approved contraceptive precautions during the trial and for 3 months following the last dose of study drug. Female with child bearing potential must have had a negative serum pregnancy test and must be non-breastfeeding.
9. Provide written informed consent voluntarily.

Exclusion Criteria:

1. Prior treatment with selective FGF19-FGFR4 inhibitor and / or treatment with Pan FGFR inhibitor.
2. Received any anti-tumor treatment within 4 weeks before the first use of the study drug.
3. Treatment with surgery, COVID-19 vaccine, or investigational drug within 4 weeks prior to the first study treatment administration.
4. CYP3A4 strong inducer used within 14 days prior to the first administration or required during the study, or CYP3A4 strong inhibitor have used within 1 week before the first study treatment administration; or CYP3A4 strong inhibitor and P-gp, BCRP transporter strong inhibitor have to be used during the study.
5. Patients with any ≥Grade 1 toxicity (as per NCI CTC AE Version 5.0) related to prior anti-cancer therapy.
6. Other malignant tumors requiring any active treatment at the same time.
7. CNS metastases that are untreated or symptomatic or uncontrolled, so it is not suitable to be included in the group according to the judgment of the investigator.
8. Pleural/peritoneal fluid or pericardial effusion with clinical signs or requiring symptomatic management.
9. Active infection and need systemic anti infection treatment within 7 days before the first use of the study drug.
10. History of autoimmune diseases and immunodeficiency, including HIV positive test, or have other acquired and congenital immunodeficiency diseases, or have a history of organ transplantation.
11. Active hepatitis B, hepatitis C virus infection.
12. History of uncontrollable or serious cardiovascular and cerebrovascular diseases.
13. Unable to swallow drugs orally, or there are conditions that seriously affect gastrointestinal absorption as judged by the investigator.
14. Symptomatic irritable bowel syndrome and requires treatment.
15. Known alcohol or drug dependence.
16. Mental disorders or poor compliance.
17. The investigator believes that the patients are not suitable for this clinical study due to other reasons.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose(MTD) | At the end of Cycle 1 (each cycle is 28 days)
  Maximum tolerated dose
Overall Response Rate (ORR) in stage 2 | up to approximately 2 years
  Overall Response Rate

SECONDARY OUTCOMES:
Occurrence and frequency of adverse events (AE) and serious adverse events (SAE) | 12 months
  Rate of adverse events (AE) and serious adverse events (SAE)
Overall Response Rate (ORR) in stage 1 | 12 months
  Overall Response Rate
Duration of Response (DOR) | 12 months
  Duration of Response
Disease Control Rate (DCR) | 12 months
  Disease Control Rate
Progression-Free Survival (PFS) | 12 months
  Progression-free survival
Overall Survival (OS) | 12 months
  Overall Survival
Pharmacokinetic profile,e.g.AUC of SYHX2005 | 12 months
  Area Under the Plasma Concentration Versus Time Curve (AUC)